CLINICAL TRIAL: NCT03028415
Title: A Multi-Center, Randomized, Pivotal Study Evaluating AMPLEX Compared To Autogenous Bone Graft in Subjects Indicated for Arthrodesis Surgery Involving the Hindfoot or Ankle
Brief Title: AMPLEX Ankle Fusion and Hindfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000226; G150153 (Other: IDE Number)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-08

CONDITIONS: Arthrodesis Surgery Involving the Hindfoot or Ankle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- AMPLEX (Experimental)
  Interventions: Device: AMPLEX
- Autogenous Bone Graft (ABG) (Active Comparator)
  Interventions: Procedure: Autogenous Bone Graft (ABG)

INTERVENTIONS:
Device: AMPLEX — A bone graft substitute
  Arms: AMPLEX
Procedure: Autogenous Bone Graft (ABG) — Control material administered by surgical implant
  Arms: Autogenous Bone Graft (ABG)

SUMMARY:
To demonstrate that AMPLEX is non-inferior to autogenous bone graft (ABG) for bone fusion in a population indicated for single, double, or triple hindfoot arthrodesis or ankle arthrodesis surgery with supplemental graft material.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Indicated for ankle or hindfoot arthrodesis and require one of the following arthrodesis procedures:

Tibiotalar (ankle); Talocalcaneal (subtalar); Talonavicular; Calcaneocuboid; Double hindfoot (e.g., talonavicular and talocalcaneal joints); Triple hindfoot (subtalar, talonavicular and calcaneocuboid joints)

* Presents with pain on weight-bearing of at least 40 mm on a 100 mm VAS at the area indicated for arthrodesis
* Presents with at least one comorbid risk factors that warrant the use of supplemental autogenous bone or allograft:

Radiographic evidence of bone defect, deficit, subsidence or subchondral cyst; More than one joint to be fused; Involvement of other adjacent or nonadjacent joints; Large surface area; Intra-articular or extra-articular deformity; Post-traumatic arthritis; Diagnosis of osteoporosis

* The Investigator determines if the joint space(s) can be adequately filled with graft material (AMPLEX or ABG) according to the following parameters:

Single hindfoot joint fusion: up to 5 cm^3; Double or triple hindfoot fusion: each individual joint up to 5 cm^3, but overall, not more than 10 cm3 for the full complement of joints; Ankle fusion: up to 10 cm^3

* Each fused joint can be rigidly stabilized with with at least 1 and no more than 3 screws across the fusion plane. (Supplemental pins and staples may be used, as well as supplemental screws and plates external to the fusion site(s))
* Willing and able to comply with all study requirements including all postoperative clinical and radiographic evaluations
* For women of childbearing potential (not post-menopausal for 12 months or surgically sterile), a urine pregnancy test with a negative result must be obtained at screening and within 24 hours prior to procedure. These trial participants must commit to adequate birth control (e.g., oral contraceptive, two methods of barrier birth control, or abstinence) through the 78 week follow-up

Exclusion Criteria:

* Bone deficit requiring a structural graft
* Charcot foot disease
* Radiographic evidence of open physes
* Prior arthroplasty, arthrodesis, major surgical repair or reconstruction of the index ankle or hindfoot joint(s)
* Requires osteotomy or fusion of the midfoot joints
* BMI greater than 45 kg/m^2
* Documented medical history of, or radiographic evidence of, a bone disease (e.g. avascular necrosis) or other condition (e.g., osteolysis) that would preclude the subject from receiving screw fixation in the opinion of the surgeon
* Requires intramedullary nail fixation or an external fixator
* Comorbidity that would limit the ability to administer any functional measurements such as FAAM-ADL
* Has at the time of surgery, a systemic infection or local infection at the site of surgery
* Medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival or interfere with ambulation or rehabilitation (e.g., history of transient ischemic attack, stroke or liver disease)
* HgbA1c level greater than or equal to 8%
* Known hypersensitivity to any of the components of the product [e.g. B2A peptide, Hydroxyapatite (HA): beta-tricalcium phosphate (βTCP), ceramic granule]
* Currently receiving treatment with a drug known to interfere with bone metabolism [e.g., systemic corticosteroid therapy (topical corticosteroid therapy is permissible), methotrexate]
* Has previously received treatment with a drug known to interfere with bone metabolism [e.g., systemic corticosteroid therapy (topical corticosteroid therapy is permissible), methotrexate] and in the opinion of the investigator could continue to negatively interfere with bone metabolism or bone healing
* History of any severe allergy or anaphylaxis, or a history of hypersensitivity to protein pharmaceuticals [e.g., monoclonal antibodies or gamma globulins, recombinant Bone Morphogenetic Proteins (BMPs)]
* Medical condition requiring radiation, chemotherapy or immunosuppression
* Have a prior or active history of malignancy (except for basal cell carcinoma of the skin)
* Has a history of autoimmune disease known to affect bone metabolism. Examples include spondyloarthropathies (e.g., ankylosing spondylitis, Crohn's disease, and ulcerative colitis), Juvenile Arthritis, Grave's disease and Hashimoto's thyroiditis; Rheumatoid Arthritis is allowed
* Have pathological or genetic liver disease or who have clinically significant, elevated baseline liver function enzymes
* Has obvious and/or documented alcohol or illicit drug addictions
* Is a prisoner in a correctional institution/facility
* Actively involved in litigation or workman's compensation
* Has participated in clinical studies evaluating investigational devices, pharmaceuticals or biologics within 6 months of randomization
* Requires chronic therapeutic use of NSAID during the first 6 post-operative weeks (except aspirin up to 325 mg bid for cardiovascular protection and/or DVT prophylaxis)
* Has previously been treated with, or exposed to, therapeutic levels of synthetic or recombinant BMPs
* Requires chronic subcutaneous or intravenous heparin therapies

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (36):
- United States (28):
  - Physician Research Group, Gilbert, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - California Pacific Orthopaedics, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Andrews Orthopaedic and Sports Medicine Center, Gulf Breeze, Florida
  - Emory Orthopaedic and Spine Hospital, Atlanta, Georgia
  - Midwest Orthopedics at Rush, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Sinai Hospital of Baltimore, Inc / Rubin Institute for Advanced Orthopedics, Baltimore, Maryland
  - Medstar, Baltimore, Maryland
  - Orthopaedic Associates of Michigan, Research and Education Institute, Grand Rapids, Michigan
  - Michigan Orthopedic Center, Lansing, Michigan
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers, Newark, New Jersey
  - University of Rochester School of Medicine, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Reconstructive Orthopaedic Associates, Philadelphia, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Campbell Clinic Orthopaedics, Germantown, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (8):
  - University of Alberta System, Edmonton, Alberta
  - Central Alberta Orthopedics, Red Deer, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - University of Laval, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 19 sites (14 sites in the United States and 5 sites in Canada) between July 2017 to July 2020.
Pre-assignment Details: A total of 80 subjects were screened in the trial, of which, 56 subjects were randomized. All the 56 randomized subjects were exposed to graft material: 39 subjects were exposed to AMPLEX and 17 subjects were exposed to autogenous bone graft (ABG).
Period: Overall Study
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Started | 39 | 17
Modified Intention-to-treat (mITT) Population | 39 | 17
Completed | 31 | 14
Not Completed | 8 | 3
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discontinued due to COVID-19 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG) | Total
Number analyzed (Participants) | 39 | 17 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.0) | 50.5 (14.4) | 53.9 (12.8)
Age, Customized [Number; unit: participants]
  <65 years | 29 | 14 | 43
  >=65 years | 10 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 21 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 39 | 16 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 36 | 12 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 10 | 29
  Canada | 20 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Met All Five Criteria for Subject Performance Composite (SPC) Endpoint
Description: Proportion of subjects who met all the following criteria for the SPC endpoint at 52 weeks: 1. Improvement in pain on weight-bearing at fusion site (≥20 mm reduction from baseline on 100 mm visual analog scale [VAS]); 2. Absence of significant graft harvest site pain (<20 mm on 100 mm VAS); 3. Improvement in Foot and Ankle Ability Measure Activities of Daily Living subscale (FAAM-ADL) (≥8 points improvement from baseline); 4. Absence of device related or procedure related serious adverse events (up to week 52); 5. Absence of secondary surgical or nonsurgical interventions intended to promote fusion (up to week 52).
  The last observation carried forward was used for subjects with missing response status at 52 weeks.
Time Frame: At week 52
Population: The mITT analysis set comprised all randomized subjects who had an attempted fusion of the index joint(s). Subjects were analyzed according to randomized (planned) treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 39 | 17
percentage of subjects | 79.5 | 35.3

2. Secondary Outcome: Proportion of Subjects Achieving Computerized Tomography (CT) Radiographic Fusion Success
Description: Defined as ≥50% bone bridging across the joint space for the full complement of joints in the absence of secondary surgical or nonsurgical interventions intended to promote fusion.
  The last observation carried forward was used for subjects with missing response status at 52 weeks.
Time Frame: At week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 39 | 17
percentage of subjects | 66.7 | 82.4

3. Secondary Outcome: Proportion of Subjects Achieving CT Radiographic Fusion Success
Description: Defined as ≥50% bone bridging across the joint space for the full complement of joints in the absence of secondary surgical or nonsurgical interventions intended to promote fusion.
Time Frame: At week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 38 | 17
percentage of subjects | 47.4 | 58.8

4. Secondary Outcome: Proportion of Subjects Achieving CT Radiographic Fusion Success
Description: as for outcome 3
Time Frame: At week 24
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 37 | 16
percentage of subjects | 73.0 | 75.0

5. Secondary Outcome: Proportion of Subjects With Change From Baseline in Pain on Weight-bearing at Fusion Site (>20 mm Reduction From Baseline on 100 mm VAS)
Description: Weight-bearing pain at the fusion site was assessed using a 100 mm visual analog scale (VAS), a subject self-assessment questionnaire. Subjects were asked to mark the location on a 100 mm line corresponding to the amount of pain they experienced, with 0 mm being "no pain" and 100 mm being "the worst pain imaginable".
  Improvement in pain on weight-bearing at the fusion site was defined as ≥ 20 mm reduction from baseline on 100 mm VAS, and is presented for this outcome measure.
Time Frame: Baseline, and at week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 37 | 16
percentage of subjects | 78.4 | 68.8

6. Secondary Outcome: Proportion of Subjects With Change From Baseline in Pain on Weight-bearing at Fusion Site (>20 mm Reduction From Baseline on 100 mm VAS)
Description: as for outcome 5
Time Frame: Baseline, and at week 24
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 36 | 16
percentage of subjects | 88.9 | 62.5

7. Secondary Outcome: Proportion of Subjects With Change From Baseline in Pain on Weight-bearing at Fusion Site (>20 mm Reduction From Baseline on 100 mm VAS)
Description: as for outcome 5
Time Frame: Baseline, and at week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 32 | 15
percentage of subjects | 90.6 | 80.0

8. Secondary Outcome: Proportion of Subjects With Absence of Graft Harvest Site Pain (<20 mm on 100 mm VAS)
Description: Graft harvest site pain was assessed using a 100 mm visual analog scale (VAS), a subject self-assessment questionnaire, and was only assessed among subjects in the ABG group. Subjects in the ABG group were asked to mark the location on a 100 mm line corresponding to the amount of pain they experienced with 0 mm being "no pain" and 100 mm being "the worst pain imaginable".
  Absence of significant graft harvest site pain was defined as <20 mm on 100 mm VAS, and is presented for this outcome measure.
Time Frame: At week 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 15
percentage of subjects | 33.3

9. Secondary Outcome: Proportion of Subjects With Absence of Graft Harvest Site Pain (<20 mm on 100 mm VAS)
Description: as for outcome 8
Time Frame: At week 6
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 15
percentage of subjects | 60.0

10. Secondary Outcome: Proportion of Subjects With Absence of Graft Harvest Site Pain (<20 mm on 100 mm VAS)
Description: as for outcome 8
Time Frame: At week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 15
percentage of subjects | 73.3

11. Secondary Outcome: Proportion of Subjects With Absence of Graft Harvest Site Pain (<20 mm on 100 mm VAS)
Description: as for outcome 8
Time Frame: At week 24
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 15
percentage of subjects | 60.0

12. Secondary Outcome: Proportion of Subjects With Absence of Graft Harvest Site Pain (<20 mm on 100 mm VAS)
Description: as for outcome 8
Time Frame: At week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 16
percentage of subjects | 68.8

13. Secondary Outcome: Change From Baseline in FAAM-ADL
Description: Functional improvement was assessed using the Foot and Ankle Ability Measure Activities of Daily Living (FAAM-ADL) subscale, a subject self-assessment questionnaire that consists of 21 items pertaining to basic functional activities. Each item is scored on a 5 point Likert scale anchored by 4 (no difficulty at all) and 0 (unable to do). The total item subscale score ranges from 0 to 84, which are transformed to a scale of 0 to 100 as the final score. Higher scores represent a higher level of function, with 100 representing no dysfunction.
Time Frame: Baseline, and at week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 37 | 16
score on a scale | 11.16 (27.67) | 7.17 (20.46)

14. Secondary Outcome: Change From Baseline in FAAM-ADL
Description: Functional improvement was assessed using the e Foot and Ankle Ability Measure Activities of Daily Living (FAAM-ADL) subscale, a subject self-assessment questionnaire that consists of 21 items pertaining to basic functional activities. Each item is scored on a 5 point Likert scale anchored by 4 (no difficulty at all) and 0 (unable to do). The total item subscale score ranges from 0 to 84, which are transformed to a scale of 0 to 100 as the final score. Higher scores represent a higher level of function, with 100 representing no dysfunction.
Time Frame: Baseline, and at week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 36 | 16
score on a scale | 25.36 (23.82) | 13.28 (17.30)

15. Secondary Outcome: Change From Baseline in FAAM-ADL
Description: as for outcome 13
Time Frame: Baseline, and at week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 32 | 15
score on a scale | 34.99 (21.51) | 11.37 (21.49)

16. Secondary Outcome: Subject Performance Composite (SPC) Endpoint
Description: Proportion of subjects who met all the following criteria for the Subject Performance Composite (SPC) endpoint at 12 weeks: 1. Improvement in pain on weight-bearing at fusion site (≥20 mm reduction from baseline on 100 mm visual analog scale [VAS]); 2. Absence of significant graft harvest site pain (<20 mm on 100 mm VAS); 3. Improvement in Foot and Ankle Ability Measure Activities of Daily Living subscale (FAAM-ADL) (≥8 points improvement from baseline); 4. Absence of device related or procedure related serious adverse events (up to week 12); 5. Absence of secondary surgical or nonsurgical interventions intended to promote fusion (up to week 12).
Time Frame: At week 12
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 37 | 16
percentage of subjects | 40.5 | 31.3

17. Secondary Outcome: Subject Performance Composite (SPC) Endpoint
Description: Proportion of subjects who met all the following criteria for the SPC endpoint at 24 weeks: 1. Improvement in pain on weight-bearing at fusion site (≥20 mm reduction from baseline on 100 mm visual analog scale [VAS]); 2. Absence of significant graft harvest site pain (<20 mm on 100 mm VAS); 3. Improvement in Foot and Ankle Ability Measure Activities of Daily Living subscale (FAAM-ADL) (≥8 points improvement from baseline); 4. Absence of device related or procedure related serious adverse events (up to week 24); 5. Absence of secondary surgical or nonsurgical interventions intended to promote fusion (up to week 24).
Time Frame: At week 24
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 36 | 15
percentage of subjects | 66.7 | 6.7

18. Secondary Outcome: Change From Baseline in Short Form-12 (SF-12)
Description: The Short Form-12 (SF-12) Health Survey includes 12 questions from the SF-36 Health Survey. These include: 2 questions concerning physical functioning; 2 questions on role limitations because of physical health problems; 1 question on bodily pain; 1 question on general health perceptions; 1 question on vitality (energy/fatigue); 1 question on social functioning; 2 questions on role limitations because of emotional problems; and 2 questions on general mental health (psychological distress and psychological well-being). These eight domain scales were used to derive Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. All scores were calculated through scoring software. Domain scales and component summary scores ranged from 0 to 100, with a higher score considered better.
Time Frame: Baseline, and at week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 36 | 16
score on a scale
  SF-12 Physical component summary (Week 24) | 9.1 (11.2) | 5.3 (7.1)
  SF-12 Mental component summary (Week 24) | 2.0 (12.5) | -3.6 (9.2)

19. Secondary Outcome: Change From Baseline in Short Form-12 (SF-12)
Description: as for outcome 18
Time Frame: Baseline, and at week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
Number analyzed (Participants) | 32 | 15
score on a scale
  SF-12 Physical component summary (Week 52) | 10.5 (10.7) | 3.8 (7.4)
  SF-12 Mental component summary (Week 52) | 4.4 (11.6) | -0.8 (11.0)

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent up to 78 weeks
Description: A treatment-emergent AE was any AE occurring after the initiation of the surgery. If the timing of an AE could not be established in relation to the initiation of the surgery, it was considered as a treatment-emergent AE. Only treatment-emergent AEs are presented.
Arm/Group | AMPLEX | Autogenous Bone Graft (ABG)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/17
Serious Adverse Events (participants affected / at risk) | 7/39 | 7/17
Other Adverse Events (participants affected / at risk) | 27/39 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMPLEX (N=39) | Autogenous Bone Graft (ABG) (N=17)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMPLEX (N=39) | Autogenous Bone Graft (ABG) (N=17)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Implant site irritation (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (3) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03028415/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03028415/SAP_001.pdf